CLINICAL TRIAL: NCT07282977
Title: Efficacy of Three Gingival Displacement Methods: A Randomized Clinical Trial
Brief Title: Efficacy of Three Gingival Displacement Methods
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanPPH
Record Dates: First submitted 2025-11-24; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Tooth Defect; Teeth Restoration
Keywords: gingival displacement; gingival retraction; gingival retraction cord; gingival retraction paste; hemostatic gel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gingival retration cord (Experimental): give the patients in this group the gingival displacemet treatment with retraction cord
  Interventions: Procedure: gingival retraction cord
- gingival retraction paste (Experimental): give the patients in this group the gingival displacemet treatment with retraction paste
  Interventions: Procedure: gingival retraction paste
- gingival retration cord+ hemostatic gel (Experimental): give the patients in this group the gingival displacemet treatment with retraction cord impregnated with hemostatic gel
  Interventions: Procedure: gingival retraction cord+hemostatic gel

INTERVENTIONS:
Procedure: gingival retraction cord — After tooth preparation, the prepared abutment tooth was rinsed and dried. A preliminary impression was taken using heavy-body silicone. An appropriately sized retraction cord (Ultrapak, #000-#0) was selected and gently packed into the gingival sulcus of the prepared tooth using a cord packer. The cord was left in the gingival sulcus for 7-8 minutes. Following cord removal, light-body silicone was immediately injected around the gingival sulcus of the prepared abutment tooth and into the preliminary impression tray, followed by seating of the preliminary impression tray to obtain the final impression.
  Arms: gingival retration cord
Procedure: gingival retraction paste — After tooth preparation, the prepared abutment tooth was rinsed and dried. A preliminary impression was taken using heavy-body silicone. Retraction paste was injected into the gingival sulcus surrounding the prepared abutment tooth. The retraction paste was left in place for 2 minutes per the manufacturer's instructions, then thoroughly rinsed, and the prepared abutment tooth was air-dried. Light-body silicone was immediately injected around the gingival sulcus and into the preliminary impression tray, followed by seating of the preliminary impression tray to obtain the final impression.
  Arms: gingival retraction paste
Procedure: gingival retraction cord+hemostatic gel — Appropriately sized retraction cords (Ultrapak, sizes #000-#0) were pre-soaked in hemostatic gel prior to use. After tooth preparation, the prepared abutment tooth was rinsed and dried. A preliminary impression was taken using heavy-body silicone. The gel-soaked retraction cords were gently packed into the gingival sulcus using a cord packer. After 7-8 minutes, the cords were removed, followed by rinsing and drying of the prepared abutment tooth. Light-body silicone was immediately injected around the gingival sulcus and into the preliminary impression tray, followed by seating of the preliminary impression tray to obtain the final impression.
  Arms: gingival retration cord+ hemostatic gel

SUMMARY:
The goal of this clinical trial is to find the best gingival displacement method for taking impressions of artificial full crowns with subgingival margins. The main question it aims to answer is:

Which of the three common gingival displacement methods works best? Researchers will compare three methods: gingival retraction cord, gingival retraction paste, and gingival retraction cord + hemostatic gel, to see which is optimal.

Participants will:

Receive one of the three gingival displacement treatments during impression taking.

Fill out a VAS form to rate their pain.

DETAILED DESCRIPTION:
The success and longevity of dental protheses largely depends on the health of periodontium. To fabricate restorations with well-adapted margins, accurate impressions are imperative. Nevertheless, obtaining accurate impressions is challenging when preparations have intentionally placed cervical margins in the gingival sulcus for esthetic or functional purposes. In such cases, gingival displacement is required to ensure that impression materials can penetrate the gingival sulcus and capture the fine details of the prepared abutment margins.

Gingival displacement is the process in which the marginal gingiva is temporarily deflected by external force, and the sulcus opens to facilitate the entry of impression materials. Its objective should be to facilitate obtaining an accurate impression of the tooth preparation without damaging the periodontium. Gingival displacement techniques can be classified into mechanical, chemical, and surgical categories, or into non-surgical and surgical categories. Non-surgical methods can be alternatively classified into retraction cord methods and non-cord methods.

Traditionally, retraction cords have been widely utilized for gingival displacement. However, the retraction cord technique is associated with several drawbacks. First, the pressure exerted by retraction cords can reach up to 5000 kPa, a magnitude that exceeds the recovery capacity of the epithelial attachment, which consequently impairs the integrity of the epithelial attachment. Second, the applied mechanical force may induce bleeding and soft tissue trauma, which can potentially result in subsequent gingival recession. Third, patients frequently report significant levels of discomfort or pain during the procedure. Despite these limitations, cord methods remain the most widely used technique in clinical settings today. Moreover, to address bleeding and crevicular fluid seepage, impregnated retraction cords containing hemostatic agents, vasoconstrictors, or astringents have been introduced into clinical practice.

On the other hand, non-cord methods and materials are gaining increasing acceptance among dental practitioners, with retraction paste being a prominent example. Retraction paste has attracted considerable attention due to its distinct advantages: ease of application, shorter operation time, reduced patient discomfort, no requirement for anesthesia, facilitation of a dry operating field, and minimized tissue trauma compared to retraction cords. Unfortunately, cordless methods also have inherent limitations, such as insufficient gingival sulcus exposure.

Numerous researchers have investigated various gingival displacement methods and materials to assess their efficacy and safety. Unfortunately, study results have been inconsistent or even contradictory, and no consensus has been reached regarding the most appropriate gingival displacement methods and materials. Existing evidence demonstrates that current displacement methods fail to meet clinical requirements, which has prompted the development of new materials, and medications for this purpose. To date, no satisfactory solutions have been identified. Furthermore, high-quality randomized clinical trials (RCTs) focusing on gingival displacement remain limited. The objective of this randomized controlled clinical trial (RCT) is to evaluate the efficacy of three gingival displacement methods. The null hypothesis was that the three methods would yield equivalent displacement effects.

In the present study the enrolled Patients will get different gingival displacement treatment and fill out the VAS form. The objective of the RCT study is to see which method is optimal for gingival displacement.

ELIGIBILITY:
Inclusion Criteria:

* need for single crown restoration of maxillary anterior teeth, healthy periodontal status, and subgingival preparation margins on the buccal surface of the affected teeth.

Exclusion Criteria:

* requirement for more than one restoration, restoration in other dental quadrants, and supragingival preparation margins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
horizontal sulcus width of gingival displacement | baseline
  After tooth preparation, gingival displacement material was applied to each group and then silicone impressions were taken using the two-step impression technique, and die stone models were poured.The horizontal displacement width of the sulcus was measured on the cast, defined as the linear distance between the margin of the prepared tooth and the adjacent gingival replica on the cast. The mearsurement procedure was carried out with an optical microscope.

SECONDARY OUTCOMES:
gingival sulcus bleeding | baseline
  After the removal of gingival displacement materials, there will be gingival sulcus bleeding in some patients whereas not in other patients. In the present study, this outcome will be classified into two types: bleeding present and no bleeding present according to the bleeding status of the prepared tooth.
patient- reported pain | baseline
  Immediately after gingival displacement and impression taking, patients were asked to complete a Visual Analogue Scale (VAS) to assess their pain level during the gingival displacement procedure. The VAS scale was anchored by "no pain" (0 point) and "unbearable pain" (10 point). Patients completed the VAS independently without interference from the investigators. The scoring criteria were defined as follows: no pain to mild pain: ≤ 3 points; moderate pain (tolerable): 4-6 points; severe pain (intolerable): 7-10 points.

CONTACTS AND LOCATIONS:
Locations (1):
- department of stomatology, Henan provincial people's hospital, People's hospital Henan university., Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No